CLINICAL TRIAL: NCT02128217
Title: Sofosbuvir-Containing Regimens Without Interferon For Treatment of Acute HCV in HIV-1 Infected Individuals (SWIFT-C)
Brief Title: Sofosbuvir-Containing Regimens Without Interferon For Treatment of Acute Hepatitis C Virus (HCV) Infection
Acronym: SWIFT-C
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Advancing Clinical Therapeutics Globally for HIV/AIDS and Other Infections (Network)
Collaborators: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ACTG A5327; UM1AI068636 (NIH)
Record Dates: First submitted 2014-04-29; First posted 2014-05-01 (Estimated); Results first posted 2018-03-30 (Actual); Last update posted 2018-04-27 (Actual); Status verified 2018-03

CONDITIONS: HIV-1 Infection; Hepatitis
MeSH Terms: conditions — Hepatitis | interventions — Sofosbuvir; Ribavirin; ledipasvir, sofosbuvir drug combination

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cohort 1: SOF+weight-based RBV for 12 wks (Experimental): Participants in Cohort 1 were assigned Sofosbuvir (SOF)+weight-based ribavirin (RBV) for 12 weeks. Follow-up visits occurred through to 24 weeks after the end of treatment.
  Interventions: Drug: Sofosbuvir; Drug: Ribavirin
- Cohort 2: LDV/SOF for 8 wks (Experimental): Participants in Cohort 2 were assigned Ledipasvir/Sofosbuvir for 8 weeks. Follow-up visits occurred through to 24 weeks after the end of treatment.
  Interventions: Drug: Ledipasvir/Sofosbuvir

INTERVENTIONS:
Drug: Sofosbuvir — Participants received one 400 mg tablet of sofosbuvir (SOF) orally every morning with food
  Other Names: SOF
  Arms: Cohort 1: SOF+weight-based RBV for 12 wks
Drug: Ribavirin — Participants received weight-based ribavirin RBV orally, 2 times a day, every morning and every evening, with food. Weight under 75 kg, 600 mg (3 tablets) morning and 400 mg (2 tablets) evening. Weight over 75 kg, 600 mg (3 tablets) morning and 600 mg (3 tablets) evening. The dose of RBV was based on subject's weight at entry. Changes in weight after entry did not require a change in dose. Doses were only changed for toxicity management.
  Other Names: RBV
  Arms: Cohort 1: SOF+weight-based RBV for 12 wks
Drug: Ledipasvir/Sofosbuvir — Participants received one daily fixed-dose combination tablet orally every morning of 90 mg of Ledipasvir (LDV) and 400 mg of SOF.
  Other Names: LDV/SOF
  Arms: Cohort 2: LDV/SOF for 8 wks

SUMMARY:
Early identification of acute HCV infection is essential to prevent chronic infections and the long-term liver disease complications that may occur. Early identification and treatment of HCV during the acute phase can result in significantly higher response rates with shorter durations of therapy.

Pegylated-interferon alfa (PEG-IFN) was the typical treatment for HCV infection. Participants subcutaneously inject PEG-IFN where the average duration of treatment was approximately 20 weeks. With the advancement of direct-acting antivirals (DAAs), it was possible to see if a new DAA might be non-inferior compared to (PEG-IFN).

The study was designed to see if a fixed-dose combination tablet can replace the old HCV treatments by being more effective, safer and better tolerated in HIV-infected participants with new HCV infection. The study was a Phase I, open-label, two cohort clinical trial, in which 44 acutely HCV-infected HIV-1 positive participants were enrolled. Participants in each cohort were evaluated in two steps: on treatment (Step 1) and follow-up after discontinuing study treatment (Step 2). The cohorts were enrolled sequentially. Participants in Cohort 1 were enrolled and administered oral Sofosbuvir (SOF) in combination with weight-based ribavirin (RBV). Participants in Cohort 2 were enrolled and administered an oral fixed dose combination of Ledipasvir/Sofosbuvir (LDV/SOF).

DETAILED DESCRIPTION:
The first cohort opened with SOF/RBV treatment for 12 weeks and accrued 17 participants. All participants under Cohort 1 were to visit the clinical site at weeks 0, 1, 2, 4, 8, and 12 when on treatment (Step 1), then visit the clinical site again at 2, 4, 8, 12 and 24 weeks during follow-up after discontinuing study treatment (Step 2).

The second cohort opened for an 8-week treatment of LDV/SOF and included at least 27 subjects. All participants under Cohort 2 were to visit the clinical site at weeks 0, 1, 2, 4, and 8 when on treatment (Step 1), then visit the clinical site again at 2, 4, 8, 12 and 24 weeks during follow-up after discontinuing study treatment (Step 2).

Both cohorts were monitored for safety and HCV viral load response while the participants were on treatment.

The primary objective did not compare the cohorts together; instead, each study cohort was formally assessed for efficacy with sustained virologic response 12 weeks after treatment based on non-inferiority criteria compared to a historical SVR rate of 60% separately.

ELIGIBILITY:
A5327 Eligibility Criteria (Cohort 1 and Cohort 2)

Step 1 inclusion criteria for both cohorts (Cohort 1 and Cohort 2)

* HIV-1 infection, documented by any licensed rapid HIV test or HIV enzyme or chemiluminescence immunoassay (E/CIA) test kit at any time prior to study entry and confirmed by a licensed Western blot or a second antibody test by a method other than the initial rapid HIV and/or E/CIA, or by HIV-1 p24 antigen, or plasma HIV-1 RNA viral load. [NOTE: The term "licensed" refers to a FDA-approved kit, which is required for all IND studies.] WHO (World Health Organization) and CDC (Centers for Disease Control and Prevention) guidelines mandate that confirmation of the initial test result must use a test that is different from the one used for the initial assessment. A reactive initial rapid test should be confirmed by either another type of rapid assay or an E/CIA that is based on a different antigen preparation and/or different test principle (e.g., indirect versus competitive), or a Western blot or a plasma HIV-1 RNA viral load.
* A documented confirmation of acute HCV infection within 6 months prior to A5327 entry or HCV reinfection as described below:

  1. Acute HCV infection was defined as meeting one of the following criteria and exclusion of other causes of acute hepatitis:

     * New (<24 weeks prior to initial A5327 entry) ALT elevation to ≥5X upper limit of normal (ULN) OR >250 U/L in patients with documented normal ALT in the preceding 12 months or ≥10X ULN OR >500 U/L in patients with abnormal or no measured ALT baseline in the preceding 12 months with detectable HCV RNA excluding those with any prior positive anti-HCV. OR
     * Detectable HCV RNA with prior negative anti-HCV Ab or undetectable HCV RNA within the preceding 6 months.
  2. Acute HCV reinfection was defined by documentation of clearance of prior infection (as evidenced by positive anti-HCV Ab) either spontaneously or after treatment with two negative HCV RNA a minimum of 6 months apart AND meeting one of the following criteria in addition to exclusion of other causes of acute hepatitis:

     * New (<24 weeks prior to initial A5327 entry) ALT elevation to ≥5X ULN OR >250 U/L in patients with documented normal ALT in the preceding 12 months or ≥10X ULN OR >500 U/L in patients with abnormal or no measured ALT baseline in the preceding 12 months with detectable HCV RNA. OR
     * Positive HCV RNA with prior negative HCV RNA within the preceding 6 months.
* HCV RNA confirmed to be detectable >12 weeks after first laboratory evidence of acute HCV and still within the <24 week from first laboratory evidence of acute HCV infection window. First laboratory evidence of infection was defined as date of first elevated liver enzymes or date of first serologic evidence of HCV seroconversion and/or viremia (whichever occurs first). [NOTE: If the screening visit occurred less than 12 weeks from the first laboratory evidence of infection, then the participant was required a pre-entry study visit to confirm detectable HCV RNA at least 12 weeks from the first laboratory evidence of infection had passed. It was optimal for this pre-entry visit to occur as close as possible to 12 weeks from first laboratory evidence to ensure timely treatment. Potential participants who entered screening but who had an undetectable HCV RNA (<LLOQ TND) at the pre-entry visit (when required) exhibited evidence of possible spontaneous clearance and will not meet the entry criteria.]
* Body mass index (BMI) ≥ 18 kg/m^2
* Screening electrocardiogram (ECG) without clinically significant abnormalities as determined by the investigator.
* Willing and able to provide written informed consent.
* Men and women age ≥ 18 years.
* All participants agreed not to participate in a conception process (eg, active attempt to become pregnant or to impregnate, sperm donation, in vitro fertilization). [NOTE: Female candidates who were pregnant or breastfeeding were not eligible. A male candidate who had a pregnant female partner was not eligible for the study.]
* When participating in sexual activity that could lead to pregnancy, all participants must agree to use at least two reliable forms of contraceptive simultaneously while receiving protocol-specified medications, and for 6 months after stopping the medications. Such methods included:

  * Condoms (male or female) with or without a spermicidal agent
  * Diaphragm or cervical cap with spermicide
  * Intrauterine device (IUD)
  * Tubal ligation
  * Hormone-based contraceptive (except those containing drospirenone)

[NOTE: Providers and participants were advised that not all contraceptive choices listed above can prevent HIV transmission and that some may actually increase the risk of HIV acquisition. Study participants who were sexually active with HIV-1 negative or unknown HIV-1 serostatus partners were advised that they needed to consider effective strategies for reducing the risk of HIV transmission, as well as meeting the requirement for effective contraception during their participation in the study. Study participants discussed contraceptive choices and HIV risk reduction methods with their health care provider.]

* Participants who were not of reproductive potential (women who had been post-menopausal for at least 24 consecutive months or had undergone hysterectomy and/or bilateral oophorectomy or salpingectomy or men who had documented azoospermia or undergone vasectomy) were eligible without requiring the use of contraceptives. Acceptable documentation of sterilization and menopause was specified below.

  * Written or oral documentation communicated by clinician or clinician's staff of one of the following:
  * Physician report/letter
  * Operative report or other source documentation in the patient record (a laboratory report of azoospermia was required to document successful vasectomy)
  * Discharge summary
  * Follicle stimulating hormone-release factor (FSH) measurement elevated into the menopausal range as established by the reporting laboratory.
* Intention to comply with the dosing instructions for study drug administration and able to complete the study schedule of assessments.

Step 1 inclusion criteria for Cohort 1 only

* HIV-1 ARV therapy fell into one of the following criteria:

  1. ARV untreated, for example due to (1) lack of indication per provider (CD4 T-cell count >500 cells/mm3) or (2) decision by provider and participant to defer ARV therapy during the study drug dosing period (8 or 12 weeks), or (3) elite controller (CD4+ >200 cells/mm3). OR
  2. On a stable, protocol-approved (didanosine (ddI), stavudine (d4T), zidovudine (ZDV) excluded), ARV regimen for >8 weeks prior to screening with a CD4 T-cell count >200 cells/mm3 and a documented plasma HIV-1 RNA level <50 copies/mL or < lower limit of quantification (LLOQ) of local assay if LLOQ is >50 copies/mL by any laboratory that has a Clinical Laboratory Improvement Amendments (CLIA) certification or its equivalent ≥ 8 weeks preceding the A5327 screening visit. HIV-1 RNA levels should be within 1 year of the screening visit. Screening HIV-1 RNA must be < 50 copies/mL as measured by any local laboratory using an FDA-approved assay.
* Candidates must have had the following laboratory parameters within 10-42 days prior to study entry:

  1. Hemoglobin ≥ 12 g/dL for male, ≥11 g/dL for female participants
  2. International normalized ratio (INR) ≤1.5 x ULN unless participant was known hemophilia or was stable on an anticoagulant regimen affecting INR
  3. Albumin ≥ 3 g/dL
  4. Creatinine clearance (CrCl) ≥ 60 mL/min, as calculated by the Cockcroft-Gault equation (refer to section 6.3.5 for calculator utility link)
* Female participants of reproductive potential (defined as women who have not been post-menopausal for at least 24 consecutive months, ie, who have had menses within the preceding 24 months, or women who had not undergone surgical sterilization, specifically hysterectomy and/or bilateral oophorectomy or bilateral salpingectomy) must had a negative serum pregnancy test with a sensitivity of at least 25 mIU/mL performed during screening, within 48 hours prior to study entry.

Step 1 inclusion criteria for Cohort 2 only

* HCV genotype 1a, 1b, or 4 infection with source documentation from a CLIA-approved laboratory (or its equivalent). [NOTE: Those with mixed 1a/b genotype were classified as 1a.]
* HIV-1 ARV therapy fell into one of the following criteria:

  1. ARV untreated, for example due to (1) lack of indication per provider (CD4 T-cell count >500 cells/mm3) or (2) decision by provider and participant to defer ARV therapy during the study drug dosing period (8 or 12 weeks), or (3) elite controller (CD4+ >200 cells/mm3). OR
  2. On a stable, protocol-approved ARV regimen (the following ARVs are not allowed: ddI, d4T, and TPV/r) for >8 weeks prior to screening with a CD4 T-cell count >200 cells/mm3 and a documented plasma HIV-1 RNA level <50 copies/mL or <LLOQ of local assay if LLOQ is >50 copies/mL by any laboratory that had a Clinical Laboratory Improvement Amendments (CLIA) certification or its equivalent ≥ 8 weeks preceding the A5327 screening visit. HIV-1 RNA levels should be within 1 year of the screening visit. Screening HIV-1 RNA must be <50 copies/mL as measured by any local laboratory using an FDA-approved assay.
* Candidates must have had the following laboratory parameters within 10-42 days prior to study entry:

  1. Hemoglobin ≥9 g/dL for male and female participants
  2. International normalized ratio (INR) ≤1.5 x ULN unless participant had known hemophilia or wass stable on an anticoagulant regimen affecting INR
  3. Albumin ≥3 g/dL
  4. Creatinine clearance (CrCl) ≥60 mL/min, as calculated by the Cockcroft-Gault equation (refer to section 6.3.5 for calculator utility link)
* Female participants of reproductive potential (defined as women who had not been post-menopausal for at least 24 consecutive months, ie, who had menses within the preceding 24 months, or women who had not undergone surgical sterilization, specifically hysterectomy and/or bilateral oophorectomy or bilateral salpingectomy) must had a negative serum or urine pregnancy test within 48 hours prior to study entry by any laboratory or clinic that had a CLIA certificate or its equivalent, or was using a point-of-care (POC)/CLIA-waived test. The serum, urine or POC pregnancy test must had a sensitivity of at least 25 mIU/mL.

Step 1 exclusion criteria for both cohorts (Cohort 1 and Cohort 2)

* Received investigational drug or device within 60 days prior to study entry.
* Chronic liver disease of a non-HCV etiology (eg, hemochromatosis, Wilson's disease, α1 antitrypsin deficiency, primary sclerosing cholangitis).
* Presence of active or acute AIDS-defining opportunistic infections within 30 days prior to study entry. [NOTE: A list of AIDS-defining opportunistic infections as defined by the CDC, can be found in Appendix B of the following document: http://www.cdc.gov/mmwr/preview/mmwrhtml/00018871.htm]
* Active, serious infection (other than HIV-1 or HCV) requiring parenteral antibiotics, antivirals, or antifungals within 30 days prior to study entry.
* Infection with hepatitis B virus (HBV) defined as HBsAg positive.
* Evidence of acute hepatitis A infection defined as HAV IGM positive.
* Chronic use of systemically administered immunosuppressive agents (eg, prednisone equivalent > 10 mg/day).
* History of solid organ transplantation.
* Current or prior history of clinical hepatic decompensation (eg, ascites, encephalopathy or variceal hemorrhage).
* History of a gastrointestinal disorder (or post operative condition) that could interfere with the absorption of the study drug.
* History of significant or symptomatic pulmonary disease, cardiac disease, or porphyria.
* History of difficulty with blood collection and/or poor venous access for the purposes of phlebotomy.
* History of clinically significant illness or any other major medical disorder that may interfere with participant treatment, assessment, or compliance with study requirements, which may included active drug or alcohol use or dependence.
* Use of any prohibited concomitant medications within 30 days prior to study entry.
* Acute HIV infection defined as the phase immediately following infection during which anti-HIV antibodies are undetectable. [NOTE: Participants with early infection, defined as within the first 6 months of infection and with a positive HIV antibody, should be discussed with the A5327 protocol core team. These participants may be considered for inclusion in the study on a case by case basis with the specific documented approval of the protocol chairs.]

Step 1 exclusion criteria for Cohort 1 only

* Prior exposure to a direct-acting antiviral (DAA) targeting the HCV NS5B polymerase. [NOTE: DAAs include but are not limited to: mericitabine, ABT-333, ABT-072, BI-207127, BMS-791325, VX-222, tegobuvir, IDX719, setrobuvir, GS-9669, VX-135.]
* History of clinically significant hemoglobinopathy (eg, sickle cell disease, thalassemia).
* Known hypersensitivity to RBV, SOF, its metabolites, or formulation excipients or any other contraindication to the use of RBV or SOF.
* Currently receiving ZDV, ddI, or d4T.

Step 1 Exclusion criteria for Cohort 2 only

* Any preceding attempt at HCV treatment during this acute HCV infection episode, ie, 24 weeks prior to entry.
* Known hypersensitivity to SOF or LDV, the metabolites, or formulation excipients or any other contraindication to the use of SOF or LDV.
* Currently receiving TPV/r, ddI, d4T or amiodarone.
* Pregnancy or Breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Actual)
Dates: Start 2014-05-30 (Actual); Primary Completion 2017-02-28 (Actual); Study Completion 2017-05-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Raymond T Chung, M.D., Study Chair — Massachusetts General Hospital; Susanna Naggie, M.D., Study Chair — Duke University
Locations (12):
- United States (12):
  - 701 University of California, San Diego AntiViral Research Center CRS, San Diego, California
  - 801 University of California, San Francisco HIV/AIDS CRS, San Francisco, California
  - Whitman Walker Health CRS (31791), Washington D.C., District of Columbia
  - 2701 Northwestern University CRS, Chicago, Illinois
  - Rush Univ. Med. Ctr. ACTG CRS (2702), Chicago, Illinois
  - 101 Massachusetts General Hospital (MGH) CRS, Boston, Massachusetts
  - 7804 Weill Cornell Chelsea CRS, New York, New York
  - 7803 Weill Cornell Upton CRS, New York, New York
  - 2401 Cincinnati CRS, Cincinnati, Ohio
  - 6201 Penn Therapeutics CRS, Philadelphia, Pennsylvania
  - 31443 Trinity Health and Wellness Center CRS, Dallas, Texas
  - 31473 Houston AIDS Research Team (HART) CRS, Houston, Texas

REFERENCES:
- [Derived] Naggie S, Fierer DS, Hughes MD, Kim AY, Luetkemeyer A, Vu V, Roa J, Rwema S, Brainard DM, McHutchison JG, Peters MG, Kiser JJ, Marks KM, Chung RT; Acquired Immunodeficiency Syndrome Clinical Trials Group (ACTG) A5327 Study Team. Ledipasvir/Sofosbuvir for 8 Weeks to Treat Acute Hepatitis C Virus Infections in Men With Human Immunodeficiency Virus Infections: Sofosbuvir-Containing Regimens Without Interferon for Treatment of Acute HCV in HIV-1 Infected Individuals. Clin Infect Dis. 2019 Jul 18;69(3):514-522. doi: 10.1093/cid/ciy913. PMID 31220220
- [Derived] Naggie S, Marks KM, Hughes M, Fierer DS, Macbrayne C, Kim A, Hollabaugh K, Roa J, Symonds B, Brainard DM, McHutchison JG, Peters MG, Kiser JJ, Chung R; AIDS Clinical Trials Group (ACTG) A5327 Study Team. Sofosbuvir Plus Ribavirin Without Interferon for Treatment of Acute Hepatitis C Virus Infection in HIV-1-Infected Individuals: SWIFT-C. Clin Infect Dis. 2017 Apr 15;64(8):1035-1042. doi: 10.1093/cid/cix025. PMID 28329053
- See also: The Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 2.0, November 2014 — http://rsc.tech-res.com/docs/default-source/safety/daids_ae_grading_table_v2_nov2014.pdf
- See also: Aids Clinical Trial Group Network — http://actgnetwork.org/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 12 different study sites in the United States. For Cohort 1, the first participant enrolled on 30 May 2014; the last participant enrolled on 7 October 2014. For Cohort 2, the first participant enrolled on 31 August 2015; the last participant enrolled on 27 September 2015.
Groups:
- Cohort 1: SOF+Weight-based RBV for 12 Wks: Follow-up occurred through to 24 weeks after the end of treatment.
  Sofosbuvir (SOF): Participants received one 400 mg tablet of sofosbuvir orally every morning with food.
  Ribavirin (RBV): Participants received weight-based RBV orally, 2 times a day, every morning and every evening, with food. Weight under 75 kg, 600 mg (3 tablets) morning and 400 mg (2 tablets) evening. Weight over 75 kg, 600 mg (3 tablets) morning and 600 mg (3 tablets) evening. The dose of RBV was based on subject's weight at entry. Changes in weight after entry did not require a change in dose. Doses were only changed for toxicity management.
- Cohort 2: LDV/SOF for 8 Wks: Follow-up occurred through to 24 weeks after the end of treatment.
  Ledipasvir/Sofosbuvir (LDV/SOF): Participants received one daily fixed-dose combination tablet orally every morning of 90 mg of LDV and 400 mg of SOF.
Period: Overall Study
Arm/Group | Cohort 1: SOF+Weight-based RBV for 12 Wks | Cohort 2: LDV/SOF for 8 Wks
Started | 17 | 27
Completed | 17 | 26
Not Completed | 0 | 1
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Participants who enrolled and started first dose of study treatment.
Groups:
- Cohort 1: SOF+Weight-based RBV for 12 Wks: Follow-up occurred through to 24 weeks after the end of treatment.
  Sofosbuvir (SOF): Participants received one 400 mg tablet of sofosbuvir orally every morning with food.
  Ribavirin(RBV): Participants received weight-based RBV orally, 2 times a day, every morning and every evening, with food. Weight under 75 kg, 600 mg (3 tablets) morning and 400 mg (2 tablets) evening. Weight over 75 kg, 600 mg (3 tablets) morning and 600 mg (3 tablets) evening. The dose of RBV was based on subject's weight at entry. Changes in weight after entry did not require a change in dose. Doses were only changed for toxicity management.
- Total: Total of all reporting groups
Arm/Group | Cohort 1: SOF+Weight-based RBV for 12 Wks | Cohort 2: LDV/SOF for 8 Wks | Total
Number analyzed (Participants) | 17 | 27 | 44
Age, Continuous [Median (Inter-Quartile Range); unit: Years] | 45 [41 to 47] | 46 [38 to 50] | 45.5 [38.5 to 49.5]
Age, Customized [Count of Participants; unit: Participants]
  Age: 20-29 years | 3 | 1 | 4
  Age: 30-39 years | 1 | 8 | 9
  Age: 40-49 years | 10 | 10 | 20
  Age: 50-59 years | 2 | 6 | 8
  Age: 60-69 years | 1 | 1 | 2
  Age: 70+ years | 0 | 1 | 1
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 17 | 27 | 44
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race/Ethnicity: White Non-Hispanic | 6 | 11 | 17
  Race/Ethnicity: Black Non-Hispanic | 0 | 5 | 5
  Race/Ethnicity: Hispanic (Regardless of Race) | 11 | 9 | 20
  Race/Ethnicity: Asian, Pacific Islander | 0 | 2 | 2
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 27 | 44
Intravenous Drug History [Count of Participants; unit: Participants]
  Never | 13 | 22 | 35
  Currently | 0 | 1 | 1
  Previously | 4 | 4 | 8
Weight [Count of Participants; unit: Participants]
  Less than 75 kg | 7 | 12 | 19
  Greater than or equal to 75 kg | 10 | 15 | 25
Type of Acute HCV Infection [Count of Participants; unit: Participants]
  New Infection | 17 | 22 | 39
  Reinfection | 0 | 5 | 5
HCV Genotype [Count of Participants; unit: Participants]
  1a | 11 | 23 | 34
  1b | 2 | 3 | 5
  1 (subtype unknown) | 2 | 0 | 2
  2b | 1 | 0 | 1
  4 | 0 | 1 | 1
  Indeterminate | 1 | 0 | 1
IL28B Genotype [Count of Participants; unit: Participants]
  CC | 4 | 16 | 20
  CT | 10 | 7 | 17
  TT | 3 | 4 | 7
HCV RNA [Median (Inter-Quartile Range); unit: IU/mL] | 2280000 [272000 to 4230000] | 1490000 [32500 to 3560000] | 1500000 [117500 to 3895000]
HCV RNA Levels [Count of Participants; unit: Participants]
  < 6 million IU/mL | 15 | 21 | 36
  >= 6 million IU/mL | 2 | 6 | 8
HIV RNA [Count of Participants; unit: Participants] — Population: One participant in Cohort 1 did not have HIV RNA results obtained at baseline.
  Participants
    number analyzed (Participants) | 16 | 27 | 43
    <50 copies/mL | 15 | 27 | 42
    >= 50 copies/mL | 1 | 0 | 1
Received HIV ARVs Prior to Study Entry [Count of Participants; unit: Participants]
  Yes | 16 | 27 | 43
  No | 1 | 0 | 1
History of Sexually Transmitted Infections [Count of Participants; unit: Participants]
  Reported History of STI Diagnosis | 8 | 11 | 19
  No History of STI Diagnosis | 9 | 16 | 25

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Sustained Virologic Response 12 (SVR12)
Description: SVR12 was defined as HCV RNA undetectable less than the lower limit of quantification, Target Not Detected (<LLOQ TND) of the assay at 12 weeks after date of last dose of study treatment.
  For both Cohort 1 and Cohort 2, the 12 week measurement used for determining SVR12 was the measurement obtained closest to 84 days (i.e. 12*7 days), within the window 79 to 112 days inclusive. If a participant did not have an HCV RNA measurement within this window, then the participant was considered as having detectable HCV RNA at 12 weeks unless the preceding and subsequent HCV RNA measurements were both undetectable (<LLOQ TND).
  A two-sided 90% confidence interval was calculated for this percentage using the Blyth-Still-Casella method.
Time Frame: At 12 weeks after date of last dose of study treatment. The duration of study treatment for Cohort 1 and Cohort 2 were 12 and 8 weeks, respectively.
Population: Participants who enrolled and started at least one dose of study treatment
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Groups:
- Cohort 1: SOF+Weight-based RBV for 12 Wks: Follow-up occurred through 24 weeks after the end of treatment.
  Sofosbuvir (SOF): Participants received one 400 mg tablet of sofosbuvir orally every morning with food.
  Ribavirin (RBV): Participants received weight-based RBV orally, 2 times a day, every morning and every evening, with food. Weight under 75 kg, 600 mg (3 tablets) morning and 400 mg (2 tablets) evening. Weight over 75 kg, 600 mg (3 tablets) morning and 600 mg (3 tablets) evening. The dose of RBV was based on subject's weight at entry. Changes in weight after entry did not require a change in dose. Doses were only changed for toxicity management.
- Cohort 2: LDV/SOF for 8 Wks: Follow-up occurred through 24 weeks after the end of treatment.
  Ledipasvir/Sofosbuvir (LDV/SOF): Participants received one daily fixed-dose combination tablet orally every morning of 90 mg of LDV and 400 mg of SOF.
Arm/Group | Cohort 1: SOF+Weight-based RBV for 12 Wks | Cohort 2: LDV/SOF for 8 Wks
Number analyzed (Participants) | 17 | 27
Percentage of participants | 58.8 [36.4 to 77.5] | 100.0 [89.9 to 100.0]

2. Primary Outcome: Percentage of Participants With an Occurrence of a Grade ≥ 2 Adverse Event, Serious AE According to ICH Criteria, or Treatment-limiting AE.
Description: Any adverse event occurring after initiation of study treatment through to 28 days after the date of last dose of study treatment was included (except that an event that was ongoing at the same grade from before start of study treatment was excluded). Adverse events consisted of Grade ≥ 2 primary diagnosis, primary sign/symptoms, and primary laboratory abnormality. It also included any serious adverse event according to ICH criteria and any treatment-limiting AE (ie, an AE reported as the reason for permanent discontinuation of study treatment).
  A two-sided 90% confidence interval was calculated for the percentage using the Blyth-Still-Casella method.
Time Frame: From initiation of study treatment to 28 days after last dose of study treatment. The duration for study treatment for Cohort 1 and Cohort 2 were 12 and 8 weeks, respectively.
Population: Participants who enrolled and started first dose of study treatment.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: SOF+Weight-based RBV for 12 Wks | Cohort 2: LDV/SOF for 8 Wks
Number analyzed (Participants) | 17 | 27
Percentage of participants | 47.1 [27.7 to 68.9] | 33.3 [20.4 to 50.0]

3. Secondary Outcome: Percentage of Participants With HCV RNA Undetectable During Study Treatment
Description: HCV RNA undetectable was defined as an HCV RNA measurement <LLOQ, TND. If there was no measurement at a scheduled time, then the participant was considered as having detectable HCV RNA at that time, unless both the preceding and succeeding measurements were undetectable.
  A two-sided 90% confidence interval was calculated for each proportion using the Blyth-Still-Casella method.
Time Frame: 1, 2, 4, 8 and, for the 12-week regimen, 12 weeks after starting study treatment.
Population: Participants who successfully enrolled and started first dose of treatment.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1: SOF+Weight-based RBV for 12 Wks | Cohort 2: LDV/SOF for 8 Wks
Number analyzed (Participants) | 17 | 27
Percentage of participants
  On-treatment Week 1 | 11.8 [3.2 to 31.1] | 18.5 [9.3 to 34.7]
  On Treatment Week 2 | 29.4 [14.0 to 50.0] | 44.4 [29.1 to 61.8]
  On-treatment Week 4 | 70.6 [50.0 to 86.6] | 81.5 [65.3 to 90.7]
  On-treatment Week 8 | 100.0 [86.0 to 100.0] | 92.6 [79.6 to 98.0]
  On-treatment Week 12 | 100.0 [86.0 to 100.0] | NA [NA to NA] — On treatment week 12 visits did not apply to Cohort 2 because Cohort 2 was assigned only 8 weeks of treatment.

4. Secondary Outcome: Percentage of Participants With HCV RNA Undetectable After End of Study Treatment
Description: HCV RNA undetectable is defined as an HCV RNA measurement <LLOQ, TND. If there was no measurement at a scheduled time, then the participant was considered as having detectable HCV RNA at that time, unless both the preceding and succeeding measurements were undetectable. This outcome measure was referred to as SVR2, SVR4, SVR8 and SVR24 where SVR means sustained virologic response.
  A two-sided 90% confidence interval was calculated for the percentage using the Blyth-Still-Casella method.
Time Frame: 2, 4, 8 and 24 weeks after last dose of study treatment. The duration of study treatment for Cohort 1 and Cohort 2 were 12 and 8 weeks, respectively.
Population: Participants who successfully enrolled and started first dose of treatment.
  Note that one participant in Cohort 2 was lost to follow-up prior to week 24 and is imputed as not having SVR24 at week 24. This participant, however, had HCV RNA < LLOQ, TND at all moments from week 4 of study treatment.
Measure: Number (90% Confidence Interval); unit: Percentage of participants
Groups:
- Cohort 1: SOF+Weight-based RBV for 12 Wks: Follow-up occurred 24 through to weeks after the end of treatment.
  Sofosbuvir (SOF): Participants received one 400 mg tablet of sofosbuvir orally every morning with food.
  Ribavirin (RBV): Participants received weight-based RBV orally, 2 times a day, every morning and every evening, with food. Weight under 75 kg, 600 mg (3 tablets) morning and 400 mg (2 tablets) evening. Weight over 75 kg, 600 mg (3 tablets) morning and 600 mg (3 tablets) evening. The dose of RBV was based on subject's weight at entry. Changes in weight after entry did not require a change in dose. Doses were only changed for toxicity management.
Arm/Group | Cohort 1: SOF+Weight-based RBV for 12 Wks | Cohort 2: LDV/SOF for 8 Wks
Number analyzed (Participants) | 17 | 27
Percentage of participants
  SVR2 | 64.7 [43.2 to 82.5] | 100.0 [89.9 to 100.0]
  SVR4 | 58.8 [36.4 to 77.5] | 96.3 [84.3 to 99.6]
  SVR8 | 58.8 [36.4 to 77.5] | 96.3 [84.3 to 99.6]
  SVR24: number analyzed (Participants) | 17 | 26
  SVR24 | 64.7 [43.2 to 82.5] | 96.3 [84.3 to 99.6]

5. Secondary Outcome: Number of Participants Who Had HCV Virologic Relapse
Description: HCV virologic relapse was defined as HCV RNA undetectable at end-of-treatment but HCV RNA quantifiable during follow-up with subsequent confirmation as quantifiable.
Time Frame: From end of study treatment through to 24 weeks after end of study treatment. The duration of study treatment for Cohort 1 and Cohort 2 were 12 and 8 weeks, respectively.
Population: Participants who successfully enrolled and started first dose of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: SOF+Weight-based RBV for 12 Wks | Cohort 2: LDV/SOF for 8 Wks
Number analyzed (Participants) | 17 | 27
Participants | 7 | 0

6. Secondary Outcome: Percentage of HCV Virologic Failure Participants That Developed SOF- or LDV-Associated Resistance Mutations
Description: Percentage of participants who developed SOF- or LDV-associated resistance mutation found within HCV Virologic Failure participants. HCV virologic failure was defined as HCV RNA undetectable at end-of-treatment but HCV RNA quantifiable during follow-up with subsequent confirmation as quantifiable.
Time Frame: At time of HCV virologic failure; any time from start of study treatment to 24 weeks after end of study treatment. Duration of study treatment for Cohort 1 and 2 were 12 and 8 weeks, respectively.
Population: Participants who observed an HCV virologic failure after successfully enrolling for first dose of treatment.
Measure: Number; unit: Percentage of participants
Groups:
- Cohort 2: LDV/SOF for 8 Wks: Follow-up through to occurred 24 weeks after the end of treatment.
  Ledipasvir/Sofosbuvir (LDV/SOF): Participants received one daily fixed-dose combination tablet orally every morning of 90 mg of LDV and 400 mg of SOF.
Arm/Group | Cohort 1: SOF+Weight-based RBV for 12 Wks | Cohort 2: LDV/SOF for 8 Wks
Number analyzed (Participants) | 7 | 0
Percentage of participants | 0.00 |

7. Secondary Outcome: Count and Percentage of Participants With an Adverse Event by Type.
Description: The adverse events considered were Grade 2 or higher adverse events (primary diagnosis, primary sign and symptom, or a primary lab), SAE according to ICH criteria, or treatment-limiting adverse events. Participants may experience more than one type of adverse event.
Time Frame: Any time from start of treatment to 28 days after date of last dose of study treatment. The duration of study treatment for Cohort 1 and Cohort 2 were 12 and 8 weeks, respectively.
Population: Participants who successfully enrolled and received first dose of treatment.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: SOF+Weight-based RBV for 12 Wks | Cohort 2: LDV/SOF for 8 Wks
Number analyzed (Participants) | 17 | 27
Participants
  Primary Diagnosis | 0 | 2
  Primary Sign/Symptom | 5 | 4
  Primary Lab | 5 | 6
  Serious Adverse Event | 0 | 1
  Treatment-Limiting Adverse Event | 0 | 0

8. Secondary Outcome: Count of Participants With HIV-1 RNA <50 Copies/mL
Description: Because all except one participant had HIV-1 RNA < 50 copies/mL, participants were categorized according to whether or not their HIV-1 RNA was <5 copies/mL at each follow-up evaluation.
Time Frame: 4 and 12 weeks after start of study treatment for Cohort 1. 4 and 8 weeks after start of study treatment for the 8-week regimen used in Cohort 2)
Population: Participants who enrolled successfully, received HIV ARV regimen at entry and started first dose of treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: SOF+Weight-based RBV for 12 Wks | Cohort 2: LDV/SOF for 8 Wks
Number analyzed (Participants) | 17 | 27
Participants
  On-treatment Week 4: ≥50 copies/mL | 0 | 0
  On-treatment Week 4: <50 copies/mL | 17 | 27
  On-treatment Week 8: number analyzed (Participants) | 0 | 23
  On-treatment Week 8: ≥50 copies/mL | 0 | 0
  On-treatment Week 8: <50 copies/mL | 0 | 23
  On-treatment Week 12: number analyzed (Participants) | 17 | 0
  On-treatment Week 12: ≥50 copies/mL | 0 | 0
  On-treatment Week 12: <50 copies/mL | 17 | 0

9. Secondary Outcome: Change in CD4+ Cell Count
Description: The change in CD4+ cell count from baseline to 12 weeks after the end of study treatment.
Time Frame: Baseline to 12 weeks after end of study treatment. Duration of study treatment for Cohort 1 and Cohort 2 were 12 and 8 weeks, respectively.
Population: Participants who successfully enrolled and recieved first dose of treatment.
Measure: Mean (Standard Deviation); unit: cells/mm^3
Arm/Group | Cohort 1: SOF+Weight-based RBV for 12 Wks | Cohort 2: LDV/SOF for 8 Wks
Number analyzed (Participants) | 16 | 24
cells/mm^3 | 11 (111) | 61 (125)

10. Secondary Outcome: Self-reported Adherence to SOF
Description: Count and percentage of participants who reported having taken all doses of SOF. This outcome measure was evaluated in Cohort 1 only.
Time Frame: 1, 2, 4, 8 and 12 weeks after starting study treatment.
Population: Participants in Cohort 1 who successfully enrolled and received first dose of SOF+weight-based RBV.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: SOF+Weight-based RBV for 12 Wks | Cohort 2: LDV/SOF for 8 Wks
Number analyzed (Participants) | 17 | 0
Participants
  Week 1 | 17 |
  Week 2: number analyzed (Participants) | 16 | 0
  Week 2 | 16 |
  Week 4: number analyzed (Participants) | 16 | 0
  Week 4 | 16 |
  Week 8 | 16 |
  Week 12: number analyzed (Participants) | 15 | 0
  Week 12 | 15 |

11. Secondary Outcome: Adherence as Measured by SOF Pill Count
Description: The count and percentage of participants who had a pill count consistent with 100% of SOF doses taken. This outcome measure was evaluated in Cohort 1 only.
Time Frame: 12 weeks after starting study treatment.
Population: Participants in Cohort 1 who successfully enrolled and received first dose of SOF+weight-based RBV.
Measure: Count of Participants; unit: Participants
Groups:
- Cohort 1: SOF+Weight-based RBV for 12 Wks: Follow-up occurred through to 24 weeks after the end of treatment.
  Ribavirin (RBV): Participants received weight-based RBV orally, 2 times a day, every morning and every evening, with food. Weight under 75 kg, 600 mg (3 tablets) morning and 400 mg (2 tablets) evening. Weight over 75 kg, 600 mg (3 tablets) morning and 600 mg (3 tablets) evening. The dose of RBV was based on subject's weight at entry. Changes in weight after entry did not require a change in dose. Doses were only changed for toxicity management.
  Sofosbuvir (SOF): Participants received one 400 mg tablet of sofosbuvir orally every morning with food.
Arm/Group | Cohort 1: SOF+Weight-based RBV for 12 Wks | Cohort 2: LDV/SOF for 8 Wks
Number analyzed (Participants) | 17 | 0
Participants
  Pill count not available | 12 |
  Pill count consistent with 100% of doses taken | 4 |
  Pill count indicates <100% of doses taken | 1 |

12. Secondary Outcome: Self-reported Adherence to RBV
Description: Count and percentage of participants who reported having taken all doses of RBV. This outcome measure was evaluated in Cohort 1 only.
Time Frame: 1, 2, 4, 8 and 12 weeks after starting study treatment.
Population: Participants in Cohort 1 who successfully enrolled and received first dose of SOF+weight-based RBV.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: SOF+Weight-based RBV for 12 Wks | Cohort 2: LDV/SOF for 8 Wks
Number analyzed (Participants) | 17 | 0
Participants
  Week 1: number analyzed (Participants) | 16 | 0
  Week 1 | 16 |
  Week 2: number analyzed (Participants) | 16 | 0
  Week 2 | 15 |
  Week 4: number analyzed (Participants) | 16 | 0
  Week 4 | 15 |
  Week 8 | 16 |
  Week 12: number analyzed (Participants) | 15 | 0
  Week 12 | 15 |

13. Secondary Outcome: Adherence as Measured by RBV Pill Count
Description: The count and percentage of participants who had a pill count consistent with 100% of RBV doses taken. This outcome measure was evaluated in Cohort 1 only.
Time Frame: 12 weeks after starting study treatment.
Population: Participants in Cohort 1 who successfully enrolled and received first dose of SOF + weight-based RBV.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: SOF+Weight-based RBV for 12 Wks | Cohort 2: LDV/SOF for 8 Wks
Number analyzed (Participants) | 17 | 0
Participants
  Pill count not available | 12 |
  Pill count consistent with 100% of doses taken | 1 |
  Pill count indicates <100% of doses taken | 4 |

14. Secondary Outcome: Self-reported Adherence to LDV/SOF
Description: Count and percentage of participants who reported having taken all doses of LDV/SOF. This outcome measure was evaluated in Cohort 2 only.
Time Frame: 1, 2, 4, and 8 weeks after starting study treatment.
Population: Participants in Cohort 2 who successfully enrolled and received first dose of LDV/SOF.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: SOF+Weight-based RBV for 12 Wks | Cohort 2: LDV/SOF for 8 Wks
Number analyzed (Participants) | 0 | 27
Participants
  Week 1: number analyzed (Participants) | 0 | 25
  Week 1 |  | 25
  Week 2: number analyzed (Participants) | 0 | 25
  Week 2 |  | 25
  Week 4 |  | 27
  Week 8: number analyzed (Participants) | 0 | 23
  Week 8 |  | 18

15. Secondary Outcome: Adherence as Measured by LDV/SOF Pill Count
Description: The count and percentage of participants who had a pill count consistent with 100% of LDV/SOF doses taken.. This outcome measure was evaluated in Cohort 2 only.
Time Frame: 8 weeks after starting study treatment.
Population: Participants in Cohort 2 who successfully enrolled and received first dose of LDV/SOF.
Measure: Count of Participants; unit: Participants
Arm/Group | Cohort 1: SOF+Weight-based RBV for 12 Wks | Cohort 2: LDV/SOF for 8 Wks
Number analyzed (Participants) | 0 | 27
Participants
  Pill count not available |  | 7
  Pill count consistent with 100% of doses taken |  | 17
  Pill count indicates <100% of doses taken |  | 3

16. Secondary Outcome: Ribavirin Concentration in Plasma
Description: Ribavirin concentration in plasma. This outcome was evaluated in Cohort 1 only.
Time Frame: 4, 8, and 12 weeks after starting study treatment.
Population: Participants in Cohort 1 who successfully enrolled and received first dose of SOF + weight-based RBV.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1: SOF+Weight-based RBV for 12 Wks | Cohort 2: LDV/SOF for 8 Wks
Number analyzed (Participants) | 17 | 0
ng/mL
  Week 4 | 1803 (45.6) |
  week 8 | 2122 (30.0) |
  Week 12: number analyzed (Participants) | 16 | 0
  Week 12 | 2013 (36.4) |

17. Secondary Outcome: Cellular Concentration of Tenofovir Diphosphate (TFV-DP)
Description: Cellular concentration of tenofovir diphosphate (TFV-DP) from dried blood spot samples.
Time Frame: Baseline (before HCV study treatment), EOT (end of trial dosing), 12 weeks after end of HCV study treatment. The duration of HCV study treatment for Cohort 1 and Cohort 2 were 12 and 8 weeks, respectively.
Population: Participants who started first dose of study treatment and also took tenofovir disoporxil fumarate (TDF) for treatment of HIV infection.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: fmol/punch
Arm/Group | Cohort 1: SOF+Weight-based RBV for 12 Wks | Cohort 2: LDV/SOF for 8 Wks
Number analyzed (Participants) | 15 | 22
fmol/punch
  Baseline: number analyzed (Participants) | 13 | 22
  Baseline | 1687 (30.7) | 1516 (36.2)
  End of treatment: number analyzed (Participants) | 13 | 20
  End of treatment | 6607 (73.8) | 26846 (49.3)
  12 Weeks after end of HCV study treatment: number analyzed (Participants) | 13 | 16
  12 Weeks after end of HCV study treatment | 2100 (36.4) | 1644 (54.6)

18. Secondary Outcome: Concentration of Tenofovir Diphosphate (TFV-DP) in Peripheral Blood Mononuclear Cells (PBMCs)
Description: Concentration of tenofovir diphosphate (TFV-DP) in peripheral blood mononuclear cells (PBMCs). This outcome is measured in Cohort 1 only.
Time Frame: Baseline (before SOF + RBV dosing), EOT (end of study treatment), 12 weeks after end of HCV study treatment.
Population: Participants in Cohort 1 who successfully enrolled and received first dose of SOF + weight-based RBV and who were also taking tenofovir disoproxil fumarate (TDF) for treatment of HIV infection.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: fmol/10^6 cells
Arm/Group | Cohort 1: SOF+Weight-based RBV for 12 Wks | Cohort 2: LDV/SOF for 8 Wks
Number analyzed (Participants) | 15 | 0
fmol/10^6 cells
  Baseline: number analyzed (Participants) | 12 | 0
  Baseline | 79 (47.9) |
  End of treatment: number analyzed (Participants) | 12 | 0
  End of treatment | 149 (91.3) |
  12 Weeks after end of HCV study treatment: number analyzed (Participants) | 11 | 0
  12 Weeks after end of HCV study treatment | 81 (54.4) |

19. Secondary Outcome: Concentration of Tenofovir (TFV) in Plasma
Description: Concentration of tenofovir (TFV) in plasma among participants who took TFV for treatment of HIV infection.
Time Frame: as for outcome 17
Population: Participants who started first dose of study treatment and also took tenofovir (TFV) for treatment of HIV infection.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Cohort 1: SOF+Weight-based RBV for 12 Wks | Cohort 2: LDV/SOF for 8 Wks
Number analyzed (Participants) | 15 | 22
ng/mL
  Baseline: number analyzed (Participants) | 14 | 19
  Baseline | 98 (62.6) | 87 (97.6)
  End of treatment: number analyzed (Participants) | 13 | 20
  End of treatment | 96 (57.2) | 155 (112.1)
  12 Weeks after end of HCV study treatment: number analyzed (Participants) | 11 | 16
  12 Weeks after end of HCV study treatment | 94 (75.7) | 76 (66.2)

ADVERSE EVENTS:
Time Frame: From study entry to 24 weeks after completing study treatment. The duration of study treatment for Cohort 1 and Cohort 2 were 12 and 8 weeks, respectively.
Description: The study protocol required reporting of all new diagnoses, signs/symptoms and laboratory events of >=Grade 2, SAEs, and all signs/symptoms and laboratory events that led to a change in treatment, regardless of grade. All signs/symptoms and laboratory results that were observed or performed as part of establishing a diagnosis were requested regardless of grade. The DAIDS AE Grading Table (V2.0) and EAE Manual (V2.0) were used. All eligible participants who initiated study treatment are included.
Groups:
- Cohort 1: SOF+Weight-based RBV for 12 Wks: Follow-up occurred 24 weeks after the end of treatment. Ribavirin: Participants received weight-based RBV orally, 2 times a day, every morning and every evening, with food. Weight under 75 kg, 600 mg (3 tablets) morning and 400 mg (2 tablets) evening. Weight over 75 kg, 600 mg (3 tablets) morning and 600 mg (3 tablets) evening. The dose of RBV was based on subject's weight at entry. Changes in weight after entry did not require a change in dose. Doses were only changed for toxicity management.
  Sofosbuvir: Participants received one 400 mg tablet of sofosbuvir orally every morning with food.
- Cohort 2: LDV/SOF for 8 Wks: Follow-up occurred 24 weeks after the end of treatment. Ledipasvir/Sofosbuvir: Participants received one daily fixed-dose combination tablet orally every morning of 90 mg of LDV and 400 mg of SOF.
Arm/Group | Cohort 1: SOF+Weight-based RBV for 12 Wks | Cohort 2: LDV/SOF for 8 Wks
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/27
Serious Adverse Events (participants affected / at risk) | 0/17 | 2/27
Other Adverse Events (participants affected / at risk) | 17/17 | 24/27
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: SOF+Weight-based RBV for 12 Wks (N=17) | Cohort 2: LDV/SOF for 8 Wks (N=27)
Coronary artery disease (Cardiac disorders) | 0 | 1
Subdural haematoma (Injury, poisoning and procedural complications) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1: SOF+Weight-based RBV for 12 Wks (N=17) | Cohort 2: LDV/SOF for 8 Wks (N=27)
Fatigue (General disorders) | 2 | 1
Pyrexia (General disorders) | 1 | 0
Genitourinary tract gonococcal infection (Infections and infestations) | 1 | 0
Alanine aminotransferase increased (Investigations) | 14 | 20
Aspartate aminotransferase increased (Investigations) | 14 | 18
Blood alkaline phosphatase abnormal (Investigations) | 0 | 2
Blood alkaline phosphatase increased (Investigations) | 1 | 2
Blood bilirubin increased (Investigations) | 3 | 5
Blood cholesterol increased (Investigations) | 2 | 0
Blood creatinine increased (Investigations) | 1 | 4
Blood glucose decreased (Investigations) | 0 | 4
Blood glucose increased (Investigations) | 2 | 3
Blood phosphorus decreased (Investigations) | 1 | 0
Blood potassium decreased (Investigations) | 0 | 2
Blood sodium decreased (Investigations) | 1 | 1
Lipase abnormal (Investigations) | 3 | 0
Lipase increased (Investigations) | 0 | 2
Low density lipoprotein increased (Investigations) | 1 | 0
Neutrophil count decreased (Investigations) | 0 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1 | 0
Headache (Nervous system disorders) | 0 | 2
Initial insomnia (Psychiatric disorders) | 1 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 1 | 1
Blister (Skin and subcutaneous tissue disorders) | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
In accordance with the Clinical Trials Agreement between NIAID (DAIDS) and company collaborators, NIAID (DAIDS) provides companies with a copy of any abstract, press release, or manuscript prior to submission for publication with sufficient time for company review and comment. The publication/other disclosure can be delayed for up to 30 additional business days for manuscripts and five (5) business days for abstracts, to preserve U.S. or foreign patent or other intellectual property rights.

DOCUMENTS (3):
  • Statistical Analysis Plan: Cohort 1 (2014-07-07): https://cdn.clinicaltrials.gov/large-docs/17/NCT02128217/SAP_000.pdf
  • Statistical Analysis Plan: Cohort 2 (2017-03-15): https://cdn.clinicaltrials.gov/large-docs/17/NCT02128217/SAP_001.pdf
  • Study Protocol (2015-07-02): https://cdn.clinicaltrials.gov/large-docs/17/NCT02128217/Prot_002.pdf